CLINICAL TRIAL: NCT07193628
Title: An Open-label, First-in-human, Dose-escalation and Dose-expansion, Phase I Study of Fully Human B7H3/IL13Ra2 Bispecific Armored Chimeric Antigen Receptor T-Cell Therapy for Treatment of Recurrent or Refractory Glioblastoma
Brief Title: B7H3/IL13Ra2 Bispecific Armored Chimeric Antigen Receptor T-Cell Therapy Study for Recurrent/Refractory Glioblastoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0424
Record Dates: First submitted 2025-09-17; First posted 2025-09-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Refractory Glioblastoma; Recurrent Glioblastoma
Keywords: refractory glioblastoma; recurrent glioblastoma; Immunotherapy, Adoptive; Receptors, Chimeric Antigen; Interleukin-13 Receptor alpha2 Subunit
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 1 Treatment Group (Experimental): 2.5 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects.
  Interventions: Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 1)
- EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 2 Treatment Group (Experimental): 5 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects.
  Interventions: Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 2)
- EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 3 Treatment Group (Experimental): 10 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects.
  Interventions: Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 3)
- EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 4 Treatment Group (Experimental): 20 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects.
  Interventions: Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 4)

INTERVENTIONS:
Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 1) — 2.5 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects weekly.
  Arms: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 1 Treatment Group
Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 2) — 5 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects weekly.
  Arms: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 2 Treatment Group
Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 3) — 10 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects weekly.
  Arms: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 3 Treatment Group
Biological: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Therapy (Dose level 4) — 20 × 10⁶ EPC-003 CAR-T cells will be administered into the Ommaya reservoir of the subjects weekly.
  Arms: EPC-003 Fully Human Anti-B7H3/IL13Ra2 Armored CAR-T Cell Dose Level 4 Treatment Group

SUMMARY:
This study is an investigator-initiated, open-label Phase I clinical trial designed to evaluate the safety and efficacy of EPC-003 fully human anti-B7H3/IL13Ra2 armored Chimeric Antigen Receptor T-Cell Therapy (CAR-T) cell injection in patients with recurrent or refractory glioblastoma.

Approximately 14 patients with relapsed or refractory glioblastoma are planned to be enrolled in this trial. During the screening period (Days -28 to -15), subjects will undergo relevant examinations or observations to confirm the disease status, treatment history, and other related information. Subjects who meet the screening criteria will be enrolled in the clinical trial to receive EPC-003 treatment. Specifically, they will receive intraventricular injection of EPC-003 via Ommaya reservoir on Day 0 (D0), Day 7 (D7), Day 14 (D14), Day 21 (D21), Day 28 (D28), and Day 35 (D35), once a week, totaling 6 administrations. All CAR-T cell infusions will be delivered via intraventricular injection.

This trial comprises two phases: the first phase is the dose-escalation phase, and the second phase is the dose-expansion phase.

DETAILED DESCRIPTION:
This study is a dose-escalation and dose-expansion trial investigating the safety and efficacy of B7H3/IL13Ra2 bispecific CAR-T cell preparation in patients with recurrent or refractory glioma.

1. Dose-escalation phase Four dose groups are set in the dose-escalation phase: 2.5×10⁶, 5×10⁶, 10×10⁶, and 20×10⁶ cells per infusion, administered once weekly for a total of 6 doses.

   Dose escalation will be implemented through a combination of accelerated titration and 3+3 design. The accelerated titration design will be applied to the first 3 dose levels (with only 1 subject enrolled per level):

   If dose-limiting toxicity (DLT) or two grade ≥2 drug-related adverse events (AEs) are observed at any accelerated titration dose level, the current dose level will be expanded to 3 subjects, and subsequent trials will automatically switch to the 3+3 design.

   When 2 out of 3 subjects in a dose group experience DLT, dose escalation will be terminated, and this dose level will be identified as the non-tolerated dose. The previous dose level will then be expanded to 3 subjects.

   During the dose-escalation process, cell infusion for the first subject in the subsequent dose group can only be performed after the last subject in the previous dose group completes the 28-day DLT observation period. Within the same dose group, cell infusion for the second subject may start after the first subject completes the 2-week preliminary safety observation. The third subject will initiate cell infusion after the second subject finishes the 2-week safety observation.
2. Dose-expansion phase The dose-expansion phase will commence enrollment after preliminary safety, tolerability, and efficacy results are obtained from the dose-escalation phase. Six patients will be enrolled at the highest tolerable dose level below the non-tolerated dose to determine the maximum tolerated dose (MTD) and the recommended phase 2 dose (RP2D).

MTD is defined as the highest tolerable dose with DLT observed in ≤1/6 subjects. RP2D will be determined based on the review of safety and efficacy data collected from the dose-escalation and dose-expansion cohorts.

During the trial, if necessary and with consensus, the CAR-T cell infusion schedule may be adjusted from once weekly to once every two weeks, or the dose and dose levels may be reduced.

ELIGIBILITY:
Inclusion Criteria:

* 1: Agree to comply with the trial treatment plan and visit schedule, voluntarily enroll in the trial, and sign the informed consent form in writing.

  2: On the day of signing the informed consent form, the subject shall be aged between 18 and 75 years inclusive, with no restriction on gender.

  3: Karnofsky Performance Status (KPS) score ≥ 60%

  4: Patients with B7H3- and/or IL13Ra2-positive recurrent or refractory glioblastoma confirmed by histopathology and/or cytology, meeting the following criteria: The positive expression rate of B7H3 > 30%; The positive expression rate of IL13RA2 > 30%; Disease progression or recurrence after standard treatment (postoperative radiotherapy combined with concurrent and adjuvant chemotherapy with temozolomide); The subject has at least one measurable lesion (based on RANO criteria, with mutually perpendicular diameters both ≥ 10mm).

  5: Expected survival time ≥ 12 weeks;

  6: Subjects must have adequate organ function, meeting the following laboratory test criteria: Bone Marrow Function: Absolute Neutrophil Count (ANC) ≥ 1.5×10⁹/L; Platelet Count (PLT) ≥ 100×10⁹/L; Absolute Lymphocyte Count ≥ 0.3×10⁹/L; Hemoglobin (HGB) ≥ 8.0 g/dL. Liver function: Serum total bilirubin (T-Bil) ≤ 1.5 × upper limit of normal (ULN); for patients without liver involvement, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × ULN; for patients with liver involvement, ALT and AST ≤ 5 × ULN; Renal function: Serum creatinine ≤ 1.6 × ULN, or creatinine clearance (Ccr) ≥ 50 mL/min (calculated according to the Cockcroft-Gault formula); Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN; activated partial thromboplastin time (APTT) ≤ 1.5 × ULN; Left ventricular ejection fraction > 50%.

  7: Male subjects with reproductive potential and female subjects of childbearing age must agree to use effective contraceptive measures from the time of signing the informed consent form until 1 year after the last administration of the trial drug. For female subjects of childbearing age, the pregnancy test result within ≤7 days before the administration of the trial drug must be negative.

Exclusion Criteria:

* 1: The lesion is located in the posterior fossa structures such as the cerebellum, pons, and medulla oblongata.

  2: Complicated with meningeal metastasis or detectable malignant tumor cells in cerebrospinal fluid.

  3: Presence of epilepsy and/or high intracranial pressure that cannot be controlled or stabilized with medication.

  4: Subjects with current comorbid other central nervous system (CNS) diseases or a history of CNS diseases within 6 months prior to screening, such as uncontrolled cerebrovascular accident, transient ischemic attack, stroke, and any other autoimmune diseases involving the central nervous system.

  5: Subjects who have been diagnosed with other malignant tumors within 5 years prior to screening, excluding adequately treated carcinoma in situ of the cervix, basal cell or squamous cell carcinoma of the skin, localized prostate cancer after radical treatment, and ductal carcinoma in situ of the breast after radical treatment.

  6: Subjects who have previously received treatment targeting B7H3/IL13Ra2.

  7: Subjects who have previously received gene therapy or cell therapy.

  8: Subjects who have a history of long-term use of immunosuppressive drugs or high-dose steroid hormones; inhaled hormones used for the treatment of chronic bronchial inflammation or asthma are not affected.

  9: Subjects who have previously received allogeneic hematopoietic stem cell transplantation; or those who are eligible for and agree to undergo autologous hematopoietic stem cell transplantation.

  10: Uncontrolled active bacterial, viral, or fungal infection.

  11: Any unstable systemic disease, including but not limited to cardiovascular diseases such as unstable angina pectoris, myocardial infarction (within 6 months before screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), severe arrhythmias requiring medication, as well as pulmonary, hepatic, renal, digestive system, or metabolic diseases.

  12: Subjects who have received oral anticoagulant therapy within 1 week prior to CAR-T cell infusion.

  13: Subjects who have received anti-tumor therapy (including chemotherapy, targeted therapy, immunotherapy, TTfield therapy, investigational trial drugs, and other anti-tumor treatments) within 4 weeks prior to cell infusion or within 5 half-lives of the drug (whichever is shorter), and/or have not recovered from toxic reactions (recovery to CTCAE Version 5.0 grade ≤ 1) (except for alopecia; peripheral neurotoxicity with grade ≤ 2 is acceptable).

  14: Subjects who have received radiotherapy within 12 weeks prior to cell infusion (those with progressive disease outside the irradiated field or those in whom pseudo-progression after radiotherapy/chemotherapy can be excluded are eligible for enrollment).

  15: Subjects who have undergone major surgery or significant traumatic injury within 4 weeks prior to informed consent, or have not recovered from the side effects of surgery, or plan to undergo major surgery during the trial period.

  16: Positive for hepatitis B surface antigen (HBsAg); positive for hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA quantitative test result above the lower limit of detection; positive for hepatitis C virus (HCV) antibody with peripheral blood HCV RNA quantitative test result above the lower limit of detection; positive for human immunodeficiency virus (HIV) antibody; subjects with active syphilis infection.

  17: Pregnant or lactating women.

  18: Investigators consider that the subject has other conditions that may affect compliance or make them unsuitable for participation in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of grade 3-4 adverse events (AEs) related to B7H3/IL13Ra2 CAR-T therapy. | 28 days after first infusion of CAR-T treatment
  The incidence of grade 3-4 adverse events (AEs) related to B7H3/IL13Ra2 CAR-T therapy assessed by the NCI Common Terminology Criteria for Adverse Events (CTCAE) v5.0 criteria .

SECONDARY OUTCOMES:
Objective response rate (ORR) within 12 months of the follow-up period | From enrollment to the end of treatment at 1 year
  Overall Response Rate (ORR) is calculated by summing the percentages of patients who achieve a complete response (CR) and those who attain a partial response (PR).
Duration of response (DOR) within 12 months of the follow-up period | From enrollment to the end of treatment at 1 year
  Duration of Response (DOR) is defined as the time from the first assessment confirming Complete Response (CR) or Partial Response (PR) of the tumor to the first assessment indicating Progressive Disease (PD) or death from any cause.
Disease control rate (DCR) within 12 months of the follow-up period | From enrollment to the end of treatment at 1 year
  Disease Control Rate (DCR) is defined as the proportion of subjects who achieve Complete Response (CR), Partial Response (PR), or Stable Disease (SD).
Progression-Free Survival (PFS) within 12 months of the follow-up period | From enrollment to the end of treatment at 1 year
  Progression-Free Survival (PFS) is defined as the time from the initiation of cell infusion to the first assessment of tumor progression or death from any cause.
Overall Survival (OS) within 12 months of the follow-up period | From enrollment to the end of treatment at 1 year
  Overall Survival (OS) is defined as the length of the time from the initiation of cell infusion until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Yan, MD & PhD, Principal Investigator — Department of Neurosurgery, the Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- the Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No